CLINICAL TRIAL: NCT00926367
Title: Two-week Study to Determine and Compare the Tolerance and Irritation Potential of Topical Antibiotic and Benzoyl Peroxide to Benzoyl Peroxide and Adapalene Topical Gel Acne Medications
Brief Title: Two-week Study to Compare the Tolerance and Irritation Potential of Two Combination Topical Gel Acne Medications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C0000-405
Record Dates: First submitted 2009-06-21; First posted 2009-06-23 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Acne Vulgaris
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Benzoyl Peroxide; Adapalene; Gels

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinidamycin/ Benzoyl Peroxide (Experimental): Once-daily applications, to the randomized side of the face either left or right, of a topical antibiotic and benzoyl peroxide (BPO).
  Interventions: Drug: Clindamycin and benzoyl peroxide
- Benzoyl peroxide and adapalene (Active Comparator): Once-daily applications, to the randomized side of the face either left or right, of benzoyl peroxide (BPO) and adapalene
  Interventions: Drug: benzoyl peroxide 2.5% and adapalene 0.1% gel

INTERVENTIONS:
Drug: Clindamycin and benzoyl peroxide — Once-daily applications, to the randomized side of the face either left or right, of a topical antibiotic and benzoyl peroxide gel. This contains a topical antibiotic and benzoyl peroxide gel.
  Other Names: Duac® Topical Gel (clindamycin and benzoyl peroxide.
  Arms: Clinidamycin/ Benzoyl Peroxide
Drug: benzoyl peroxide 2.5% and adapalene 0.1% gel — Once-daily applications, to the randomized side of the face either left or right,benzoyl peroxide and adapalene gel
  Other Names: benzoyl peroxide gel and adapalene gel
  Arms: Benzoyl peroxide and adapalene

SUMMARY:
This is a single-blind (blinded expert grader), randomized, half-face study being conducted at one clinical site. On 1 side of the face, the subject will apply 1 of the 2 test products, antibiotic and benzoyl peroxide or benzoyl peroxide and adapalene gel and the contra lateral side of the face will remain non-treated to serve as a control. Approximately 25-30 male and female healthy subjects will be randomly assigned to each product

DETAILED DESCRIPTION:
This is a single-blind (blinded expert grader), parallel group, randomized, half-face study being conducted at one clinical site. On 1 side of the face, the subject will apply 1 of the 2 test products, a topical antibiotic and benzoyl peroxide or benzoyl peroxide and adapalene and the contra lateral side of the face will remain non-treated to serve as a control. Approximately 25-30 male and female healthy subjects will be randomly assigned to each product.

The subjects will be entered into a 2-week treatment phase. The once-daily applications for the study medication will be supervised at the site, Monday through Friday of each week. Subjects will apply the study product at home on Saturdays and Sundays.

A blinded expert grader will rate comparative product tolerance on each week day (excluding Saturdays and Sundays) during the study before study product is applied.

Subject questionnaires will be completed along with collection of all adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 to 45 years of age or older, able to complete the study and comply with study instructions.
* Female subjects of childbearing potential must have a negative pregnancy test. Sexually active women of childbearing potential participating in the study must have been using a medically acceptable form of contraception
* Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol specific procedures are performed.
* Is willing to discontinue use of all facial products (other than the cleanser provided and makeup or razor and facial shave product) on the face for the 3 days before their baseline/day 0 visit and use only the provided facial products and their normal makeup or razor and facial shaving product for the duration of the study.
* Is willing to avoid sunburn, tanning, tanning beds or other excessive sun exposure. Understands that if their skin tone changes significantly during the study it will be necessary to discontinue their participation.

Exclusion Criteria:

* Male subjects that have facial beards (mustache and/or goatee is acceptable).
* Is a Type I diabetic.
* Has active or chronic skin allergies.
* Has a history of acute or chronic disease that might interfere with, or increase the risk of study participation.
* Has participated in other facial studies in the preceding 30 days or other clinical studies in preceding 14 days.
* Had skin cancer treatment in preceding 12 months.
* Has damaged skin on facial areas (eg, from sunburn, tattoos, scars).
* Had any medical procedure (eg, laser resurfacing, chemical peels, plastic surgery) to facial areas in preceding 12 months.
* Had any cosmetic procedure (eg, microdermabrasion, etc.) to facial areas within 8 weeks of the baseline visit.
* Live in the same household as currently enrolled subjects.
* Any other condition or factor the investigator or his duly assigned representative believes may affect the skin response or the interpretation of the test results.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- cyberDERM, Broomall, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical research center.
Pre-assignment Details: Panelists who met the eligibility criteria and were willing to participate in the study were required to undergo a 3-day pre-trial conditioning period where they had to stop the use of all facial products. Panelists were required to use the provided Soap Free Cleanser (SFC) for washing their face and were allowed to apply their normal makeup.
Groups:
- Duac: Once-daily applications, to the randomized side of the face either left or right, of a topical antibiotic and benzoyl peroxide
- Epiduo: Once-daily applications, to the randomized side of the face either left or right, of benzoyl peroxide and adapalene
Period: Overall Study
Arm/Group | Duac | Epiduo
Started | 25 | 27
Completed | 23 | 24
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Skin Irritation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duac | Epiduo | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 24 | 26 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Skin Erythema (Redness)
Description: Assessment of erythema as part of an evaluation of tolerance of two treatments: clindamycin and benzoyl peroxide or dapsone gel. This was done by visual assessment by an independent blinded grader using the grading scale shown below.
  Grade Description 0 None 2 Mild erythema 4 Moderate confluent erythema 6 Marked erythema with some edema 8 Marked erythema, edema, possible erosion
Time Frame: Baseline, Day 1 through Day 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
Units on a scale
  Baseline | 1.56 (0.92) | 1.89 (1.01)
  Day 1 | 2.62 (1.32) | 2.65 (0.94)
  Day 2 | 2.90 (1.23) | 2.52 (1.03)
  Day 3 | 3.08 (1.23) | 2.81 (1.02)
  Day 6 | 3.17 (1.33) | 3.13 (0.89)
  Day 7 | 3.07 (1.30) | 3.08 (1.01)
  Day 8 | 2.87 (1.24) | 2.98 (1.08)
  Day 9 | 2.78 (1.36) | 3.03 (0.99)
  Day 10 | 2.89 (1.22) | 2.94 (1.02)
  Day 13 | 2.85 (1.20) | 2.83 (1.21)
  Day 14 | 2.73 (1.20) | 2.56 (1.03)
Statistical Analysis 1: Comparison: Duac vs Epiduo; Test type: Superiority or Other; p > 0.05, Dunn's Multiple Comparisons Test; A two-tailed p≤ 0.05 was taken as the level of significance for all comparisons

2. Secondary Outcome: Skin Moisture and Hydration
Description: To assess skin moisture and hydration using transepidermal water loss (TEWL). Results are measured on a continuous scale. Higher values indicate greater water loss/ lower skin moisture levels.
  Evaporative water loss measurements provide an instrumental assessment of skin barrier function(one of the layers of the skin. Damage leads to a disruption of the barrier that is accompanied by elevated water loss rates and affects skin moisture and hydration. Higher values indicate greater water loss.
Time Frame: Baseline, Days 3, 7, and 14
Measure: Mean (Standard Deviation); unit: TEWL rates (gm/m2/hr)
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
TEWL rates (gm/m2/hr)
  Baseline | 11.50 (3.65) | 13.07 (5.06)
  Day 3 | 11.38 (2.49) | 15.85 (9.12)
  Day 7 | 14.51 (3.65) | 21.65 (8.66)
  Day 14 | 13.36 (3.33) | 19.28 (8.10)

3. Primary Outcome: Skin Dryness
Description: The amount of dryness on the left and right cheek of each panelist.
  The scale used to evaluate skin dryness is:
  Grade Description 0 None 2 Slight flaking 4 Moderate flaking/scaling 6 Marked scaling / slight fissuring 8 Severe scaling, fissuring
  Expert Grader assessments of dryness were taken prior to product application on Days 0, 1, 2, 3, 6, 7, 8, 9, 10, 13 and 14.
Time Frame: Baseline, Day 1 through Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale
  Baseline | 0.12 (0.44) | 0.07 (0.27)
  Day 1 | 0.41 (0.85) | 0.25 (0.57)
  Day 2 | 0.32 (0.83) | 0.34 (0.59)
  Day 3 | 0.46 (0.91) | 0.55 (1.15)
  Day 6 | 0.61 (1.02) | 1.73 (1.76)
  Day 7 | 0.69 (1.16) | 1.85 (2.01)
  Day 8 | 0.60 (1.13) | 1.87 (2.04)
  Day 9 | 0.73 (1.28) | 2.29 (1.99)
  Day 10 | 0.56 (1.04) | 1.49 (1.77)
  Day 13 | 0.80 (1.33) | 1.26 (1.85)
  Day 14 | 0.79 (1.04) | 1.33 (1.75)
Statistical Analysis 1: Comparison: Duac vs Epiduo; Test type: Superiority or Other; p > 0.05, Dunn's Multiple Comparisons Test — A two-tailed p≤ 0.05 was taken as the level of significance for all comparisons

4. Secondary Outcome: Skin Hydration
Description: The ability of an alternating current to flow through the stratum corneum is an indirect measure of its water content. The value recorded is expressed in microsiemens. Higher values indicate greater levels of skin hydration.
  Test results were compared to measurements from the other side of the face, which was not treated instead of referring to a normal range. A normal range does not exist for this measurement. Instead, the non-treated side of the face was used as a control to determine the normal level of skin hydration.
Time Frame: Baseline, 4 hrs. post 1st Treatment, Days 3, 7, and 14
Measure: Mean (Standard Deviation); unit: Microsiemens
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
Microsiemens
  Baseline | 378.06 (131.08) | 392.09 (162.16)
  4 hrs Post 1st Treatment | 323.47 (154.30) | 415.90 (197.57)
  Day 3 | 420.97 (122.60) | 465.25 (175.65)
  Day 7 | 385.91 (156.69) | 414.77 (154.46)
  Day 14 | 401.98 (156.08) | 418.51 (139.64)

5. Secondary Outcome: Self Assessment of Burning
Description: The amount of burning on the left and right cheek of each panelist.
  The scale used to evaluate burning is:
  Scale Description:
  (scale: 0 = none to 3 = severe)
  Subject Self Assessments of burning were taken prior to product application on Days 0, 1, 2, 3, 6, 7, 8, 9, 10, 13 and 14.
Time Frame: Baseline, Day 1 through Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Duac: Patients Once-daily applications, to the randomized side of the face either left or right, of a topical antibiotic and benzoyl peroxide
- Epiduo: Patients Once-daily applications, to the randomized side of the face either left or right, of benzoyl peroxide and adapalene
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale
  Baseline | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.04 (0.20) | 0.04 (0.19)
  Day 2 | 0.04 (0.20) | 0.04 (0.19)
  Day 3 | 0.12 (0.33) | 0.15 (0.36)
  Day 6 | 0.12 (0.33) | 0.56 (0.85)
  Day 7 | 0.17 (0.48) | 0.70 (0.87)
  Day 8 | 0.17 (0.48) | 0.50 (0.81)
  Day 9 | 0.13 (0.45) | 0.27 (0.67)
  Day 10 | 0.13 (0.45) | 0.31 (0.68)
  Day 13 | 0.08 (0.28) | 0.35 (0.75)
  Day 14 | 0.08 (0.28) | 0.19 (0.57)

6. Secondary Outcome: Self Assessment of Stinging
Description: The amount of stinging on the left and right cheek of each panelist.
  The scale used to evaluate stinging is:
  Scale Description:
  (scale: 0 = none to 3 = severe)
  Subject Self Assessments of stinging were taken prior to product application on Days 0, 1, 2, 3, 6, 7, 8, 9, 10, 13 and 14.
Time Frame: Baseline, Day 1 through Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale
  Baseline | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.08 (0.28) | 0.00 (0.00)
  Day 2 | 0.08 (0.28) | 0.00 (0.00)
  Day 3 | 0.12 (0.44) | 0.04 (0.19)
  Day 6 | 0.1 (0.4) | 0.4 (0.8)
  Day 7 | 0.17 (0.48) | 0.30 (0.67)
  Day 8 | 0.17 (0.48) | 0.35 (0.69)
  Day 9 | 0.13 (0.45) | 0.15 (0.54)
  Day 10 | 0.13 (0.45) | 0.12 (0.43)
  Day 13 | 0.13 (0.34) | 0.19 (0.57)
  Day 14 | 0.08 (0.28) | 0.12 (0.43)

7. Secondary Outcome: Self Assessment of Dryness
Description: The amount of dryness on the left and right cheek of each panelist.
  The scale used to evaluate dryness is:
  Scale Description:
  (scale: 0 = none to 3 = severe)
  Subject Self Assessments of burning were taken prior to product application on Days 0, 1, 2, 3, 6, 7, 8, 9, 10, 13 and 14.
Time Frame: Baseline, Day 1 through Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale
  Baseline | 0.24 (0.44) | 0.30 (0.54)
  Day 1 | 0.2 (0.4) | 0.19 (0.40)
  Day 2 | 0.16 (0.37) | 0.15 (0.36)
  Day 3 | 0.24 (0.44) | 0.2 (0.4)
  Day 6 | 0.48 (0.77) | 0.67 (0.96)
  Day 7 | 0.54 (0.72) | 0.70 (0.91)
  Day 8 | 0.54 (0.78) | 0.81 (1.02)
  Day 9 | 0.54 (0.78) | 0.85 (1.01)
  Day 10 | 0.50 (0.78) | 0.69 (0.88)
  Day 13 | 0.50 (0.78) | 0.73 (0.96)
  Day 14 | 0.46 (0.72) | 0.69 (1.05)

8. Secondary Outcome: Self Assessment of Texture (Roughness)
Description: The amount of roughness on the left and right cheek of each panelist.
  The scale used to evaluate roughness is:
  Scale Description:
  (scale: 0 = none to 3 = severe)
  Subject Self Assessments of burning were taken prior to product application on Days 0, 1, 2, 3, 6, 7, 8, 9, 10, 13 and 14.
Time Frame: Baseline, Day 1 through Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale
  Baseline | 0.28 (0.54) | 0.15 (0.36)
  Day 1 | 0.20 (0.50) | 0.07 (0.27)
  Day 2 | 0.16 (0.47) | 0.07 (0.27)
  Day 3 | 0.32 (0.69) | 0.07 (0.27)
  Day 6 | 0.28 (0.68) | 0.33 (0.78)
  Day 7 | 0.33 (0.76) | 0.19 (0.56)
  Day 8 | 0.25 (0.61) | 0.3 (0.7)
  Day 9 | 0.29 (0.69) | 0.15 (0.46)
  Day 10 | 0.29 (0.69) | 0.15 (0.46)
  Day 13 | 0.33 (0.70) | 0.12 (0.43)
  Day 14 | 0.29 (0.69) | 0.15 (0.46)

9. Secondary Outcome: Self Assessment of Pain
Description: The amount of pain on the left and right cheek of each panelist.
  The scale used to evaluate pain is:
  Scale Description:
  (scale: 0 = none to 3 = severe)
  Subject Self Assessments of burning were taken prior to product application on Days 0, 1, 2, 3, 6, 7, 8, 9, 10, 13 and 14.
Time Frame: Baseline, Day 1 through Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale
  Baseline | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.04 (0.20) | 0.04 (0.19)
  Day 2 | 0.04 (0.20) | 0.00 (0.00)
  Day 3 | 0.04 (0.20) | 0.00 (0.00)
  Day 6 | 0.04 (0.20) | 0.1 (0.4)
  Day 7 | 0.04 (0.20) | 0.04 (0.19)
  Day 8 | 0.04 (0.20) | 0.04 (0.20)
  Day 9 | 0.04 (0.20) | 0.00 (0.00)
  Day 10 | 0.04 (0.20) | 0.00 (0.00)
  Day 13 | 0.04 (0.20) | 0.00 (0.00)
  Day 14 | 0.04 (0.20) | 0.00 (0.00)

10. Secondary Outcome: Self Assessment of Crusting
Description: The amount of crusting on the left and right cheek of each panelist.
  The scale used to evaluate crusting is:
  Scale Description:
  (scale: 0 = none to 3 = severe)
  Subject Self Assessments of burning were taken prior to product application on Days 0, 1, 2, 3, 6, 7, 8, 9, 10, 13 and 14.
Time Frame: Baseline, Day 1 through Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale
  Baseline | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.00 (0.00) | 0.00 (0.00)
  Day 2 | 0.00 (0.00) | 0.00 (0.00)
  Day 3 | 0.00 (0.00) | 0.00 (0.00)
  Day 6 | 0.00 (0.00) | 0.07 (0.38)
  Day 7 | 0.00 (0.00) | 0.04 (0.19)
  Day 8 | 0.00 (0.00) | 0.04 (0.20)
  Day 9 | 0.00 (0.00) | 0.04 (0.20)
  Day 10 | 0.00 (0.00) | 0.04 (0.20)
  Day 13 | 0.00 (0.00) | 0.00 (0.00)
  Day 14 | 0.00 (0.00) | 0.00 (0.00)

11. Secondary Outcome: Self Assessment of Blistering
Description: The amount of blistering on the left and right cheek of each panelist.
  The scale used to evaluate blistering is:
  Scale Description:
  (scale: 0 = none to 3 = severe)
  Subject Self Assessments of burning were taken prior to product application on Days 0, 1, 2, 3, 6, 7, 8, 9, 10, 13 and 14.
Time Frame: Baseline, Day 1 through Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale
  Baseline | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.00 (0.00) | 0.00 (0.00)
  Day 2 | 0.00 (0.00) | 0.00 (0.00)
  Day 3 | 0.00 (0.00) | 0.00 (0.00)
  Day 6 | 0.00 (0.00) | 0.07 (0.38)
  Day 7 | 0.00 (0.00) | 0.04 (0.19)
  Day 8 | 0.00 (0.00) | 0.00 (0.00)
  Day 9 | 0.00 (0.00) | 0.00 (0.00)
  Day 10 | 0.00 (0.00) | 0.00 (0.00)
  Day 13 | 0.00 (0.00) | 0.00 (0.00)
  Day 14 | 0.00 (0.00) | 0.00 (0.00)

12. Secondary Outcome: Self Assessment of Oiliness
Description: The amount of oiliness on the left and right cheek of each panelist.
  The scale used to evaluate oiliness is:
  Scale Description:
  (scale: 0 = none to 3 = severe)
  Subject Self Assessments of burning were taken prior to product application on Days 0, 1, 2, 3, 6, 7, 8, 9, 10, 13 and 14.
Time Frame: Baseline, Day 1 through Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale
  Baseline | 0.12 (0.33) | 0.19 (0.40)
  Day 1 | 0.08 (0.28) | 0.11 (0.42)
  Day 2 | 0.00 (0.00) | 0.04 (0.19)
  Day 3 | 0.08 (0.28) | 0.11 (0.42)
  Day 6 | 0.04 (0.20) | 0.04 (0.19)
  Day 7 | 0.00 (0.00) | 0.07 (0.27)
  Day 8 | 0.00 (0.00) | 0.04 (0.20)
  Day 9 | 0.00 (0.00) | 0.08 (0.27)
  Day 10 | 0.00 (0.00) | 0.0 (0.2)
  Day 13 | 0.00 (0.00) | 0.12 (0.43)
  Day 14 | 0.00 (0.00) | 0.08 (0.27)

13. Secondary Outcome: Product Acceptability and Preference Questionnaire - How do You Rate the Comfort of the Skin Where You Are Currently Treating With the Study Product?
Description: The subject were presented with a questionnaire at day 14 (end of study) and was asked the following question: How do you rate the comfort of the skin where you are currently treating with the study product?
  The subject replied using the following scale:
  1. - Very Comfortable
  2. - Comfortable
  3. - Somewhat Comfortable
  4. - Somewhat Uncomfortable
  5. - Uncomfortable
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale | 2.38 (1.13) | 2.23 (1.24)

14. Secondary Outcome: Product Acceptability and Preference Questionnaire - How Compliant Were You With Applying the Study Product Each and Every Day?
Description: The subject were presented with a questionnaire at day 14 (end of study) and was asked the following question: How compliant were you with applying the study product each and every day?
  The subject replied using the following scale:
  0 - Not Compliant at all (<50%)
  1. - Mostly Compliant (50%-79%)
  2. - Very Compliant (80%-100%)
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale | 2.00 (0.00) | 2.00 (0.00)

15. Secondary Outcome: Product Acceptability and Preference Questionnaire - Did You Feel That Your Skin Was Hydrated and Moisturized While You Were on Your Study Product?
Description: The subject were presented with a questionnaire at day 14 (end of study) and was asked the following question: Did you feel that your skin was hydrated and moisturized while you were on your study product?
  The subject replied using the following scale:
  1 - Yes 0 - No
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale | 0.58 (0.50) | 0.54 (0.51)

16. Secondary Outcome: Product Acceptability and Preference Questionnaire - Was the Study Product Easy to Use With Make-up?
Description: The subject were presented with a questionnaire at day 14 (end of study) and was asked the following question: Was the study product easy to use with make-up?
  The subject replied using the following scale:
  0 - Not Applicable
  1. - Very Easy
  2. - Easy
  3. - Neutral
  4. - Difficult
  5. - Very Difficult
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale | 1.04 (1.12) | 1.46 (1.14)

17. Secondary Outcome: Product Acceptability and Preference Questionnaire - What Was Your Overall Satisfaction of the Study Product?
Description: The subject were presented with a questionnaire at day 14 (end of study) and was asked the following question: What was your overall satisfaction of the study product?
  The subject replied using the following scale:
  1. - Very Satisfied
  2. - Satisfied
  3. - Neutral
  4. - Unsatisfied
  5. - Very Unsatisfied
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale | 2.29 (1.04) | 2.46 (1.03)

18. Secondary Outcome: Product Acceptability and Preference Questionnaire - How do You Rate the Ease of Application of the Study Product?
Description: as for outcome 16
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duac | Epiduo
Number analyzed (Participants) | 25 | 27
units on a scale | 1.17 (0.38) | 1.00 (0.00)

ADVERSE EVENTS:
Time Frame: 14 days
Description: Any study product-related AEs ongoing at the end of the treatment period were followed until they resolve, the condition stabilizes, the events are otherwise explained, or the subject is lost to follow-up. In addition, all SAEs were followed until resolution as previously stated for study product-related AEs.
Arm/Group | Duac | Epiduo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 13/25 | 13/27
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duac (N=25) | Epiduo (N=27)
Headache (Nervous system disorders) | 4 (4) | 5 (5)
Irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Seaonal allergies (Infections and infestations) | 1 (1) | 0 (0)
Menstrual cramps (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Toothache (General disorders) | 2 (2) | 1 (1)
Sore throat (General disorders) | 2 (2) | 3 (3)
Earache (Infections and infestations) | 0 (0) | 3 (3)
Stitches contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scratched cornea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No